CLINICAL TRIAL: NCT03825796
Title: CPX-351 Plus Enasidenib for Relapsed Acute Myelogenous Leukemia Characterized by the IDH2 Mutation
Brief Title: CPX-351 Plus Enasidenib for Relapsed AML
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-001416; NCI-2018-02998 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2019-01-30; First posted 2019-01-31 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Recurrent Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — 2-Propanol; methanesulfonic acid; enasidenib; CPX-351; Injections; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (CPX-351, enasidenib mesylate) (Experimental): See detailed description
  Interventions: Drug: Enasidenib Mesylate; Drug: Liposome-encapsulated Daunorubicin-Cytarabine

INTERVENTIONS:
Drug: Enasidenib Mesylate — Given PO
  Other Names: 2-Methyl-1-[(4-[6-(trifluoromethyl)pyridin-2-yl]-6-{[2-(trifluoromethyl)pyridin-4-yl]amino}-1,3,5-triazin-2-yl)amino]propan-2-ol Methanesulfonate; 2-Propanol, 2-Methyl-1-((4-(6-(trifluoromethyl)-2-pyridinyl)-6-((2-(trifluoromethyl)-4-pyridinyl)amino)-1,3,5-triazin-2-yl)amino)-, Methanesulfonate (1:1); AG-221 Mesylate; CC-90007; Enasidenib Methanesulfonate; Idhifa
Drug: Liposome-encapsulated Daunorubicin-Cytarabine — Given IV
  Other Names: CPX-351; Cytarabine-Daunorubicin Liposome for Injection; Liposomal AraC-Daunorubicin CPX-351; Liposomal Cytarabine-Daunorubicin; Liposome-encapsulated Combination of Daunorubicin and Cytarabine; Vyxeos

SUMMARY:
This trial evaluates how well CPX-351 and enasidenib work in treating patients with acute myeloid leukemia characterized by IHD2 mutation. Drugs used in chemotherapy, such as CPX-351, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Enasidenib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving CPX-351 and enasidenib may work better in treating patients with acute myeloid leukemia, compared to giving only one of these therapies alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the remission rate (defined as complete remission [CR]/ CR with incomplete hematologic recovery [CRi]) of the combination of liposome-encapsulated daunorubicin-cytarabine (CPX-351) plus enasidenib mesylate (enasidenib) in adults with relapsed acute myeloid leukemia (AML) characterized by a 2-hydroxyglutarate (2-HG) producing IDH2 mutations that include IDH2^R172 and IDH2^R140.

SECONDARY OBJECTIVES:

I. To evaluate persistent severe hematologic toxicity at induction day 60 in patients with a morphologic leukemia-free state (bone marrow blasts < 5%).

II. To evaluate delayed CR/CRi with enasidenib maintenance in participants with stable disease after induction with CPX-351.

III. To estimate the rate of CR plus complete remission with partial hematologic recovery (CRp) of the combination of CPX-351 plus enasidenib.

IV. To evaluate time to return of normal hematopoiesis after induction therapy. V. To evaluate 30- and 60-day survival. VI. To evaluate CPX-351 plus enasidenib as a bridge to allogeneic hematopoietic stem cell transplantation (HSCT).

EXPLORATORY OBJECTIVES:

I. To determine the co-existing mutations that are present with the IDH2 mutation and describe those that are present in patients who achieve CR/CRi.

II. To determine the depth of molecular response to induction by minimal residual disease (MRD) using next generation sequencing.

III. To estimate the subclinical cardiotoxicity of CPX-351 as measured by troponin I, electrocardiography (ECG), and echocardiography.

OUTLINE:

INDUCTION: Patients receive liposome-encapsulated daunorubicin-cytarabine intravenously (IV) over 90 minutes on days 1, 3, and 5, and enasidenib mesylate orally (PO) on days 10-60 in the absence of disease progression or unacceptable toxicity. Patients whose bone marrow is not hypoplastic receive re-induction including liposome-encapsulated daunorubicin-cytarabine IV on days 1 and 3, and enasidenib mesylate PO on days 8-60 in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION: Participants who achieve CR/CRi may proceed directly to allogeneic HSCT or receive up to 4 cycles of consolidation. Patients < 60 years receive cytarabine twice daily (BID) on days 1, 3, and 5, and patients >= 60 years receive cytarabine IV once daily on days 1-5. Patients also receive enasidenib mesylate PO on days 6-55. Treatment repeats every 28-55 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients who maintain CR/CRi after completion of consolidation therapy undergo allogeneic HSCT at the discretion of the treating physician.

MAINTENANCE: Participants who have stable disease (not meeting criteria for progressive disease, but also not achieving CR/CRi) at day 60 receive enasidenib mesylate PO daily in the absence of disease progression or unacceptable toxicity. Routine follow-up visits will be conducted at least once every 3 months for the duration of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Bone marrow blasts >= 5% that develops after CR/CRi in patient with prior history of AML, no restriction on prior number of relapses or regimens
* AML characterized by the IDH2 gene mutation, without requirement for a particular allelic frequency
* Patients previously treated with IDH2 inhibitor can be enrolled
* At least a 3-month duration of CR/CRi prior to relapse
* Relapses after allogeneic HSCT are included with a minimum of 3 from the date of allogeneic HSCT
* Up to 1 cycle of hypomethylating agent monotherapy at time of relapse is allowed, must be discontinued at least 14 days prior to start of salvage induction
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Serum total bilirubin < 2.0 mg/dL, unless considered due to Gilbert's disease or leukemic involvement
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) < 3 times the upper limit of normal, unless considered due to leukemic involvement
* Alkaline phosphatase < 3 times the upper limit of normal, unless considered due to leukemic involvement
* Serum creatinine =< 2.0 mg/dL, or creatinine clearance > 40 mL/min based on Cockcroft-Gault glomerular filtration rate (GFR)
* Females of reproductive potential as well as fertile men and their partners who are female of reproductive potential must agree to abstain from sexual intercourse or to use two highly effective forms of contraception from the time of giving informed consent, during the study, and for four months (females and males) following the last dose of IDH inhibitor. A highly effective form of contraception is defined as hormonal oral contraceptives, injectables, patches, intrauterine devices, double-barrier method (eg, synthetic condoms, diaphragm or cervical cap with spermicidal foam, cream, or gel) or male partner sterilization

Exclusion Criteria:

* Concurrent FLT3 mutation that the treating physician deems necessary to treat with FLT3-targeted therapy; whereas, patients with FLT3-mutated AML not treated with FLT3-targeted therapy can be enrolled
* Acute promyelocytic leukemia
* Inability to swallow medications or history of gastrointestinal (GI) malabsorptive disease
* Active malignancy that would limit survival by less than two years
* New York Heart Association class III or VI
* Left ventricular ejection fraction < 40%
* History of coronary stent placement that require mandatory continuation of dual-antiplatelet therapy
* Baseline QT corrected interval based on Fridericia's formula (QTcF) interval > 450 ms
* History of Wilson's disease or other copper handling disorders
* Hypersensitivity to cytarabine, daunorubicin, or liposomal products
* Active invasive fungal infection
* Active bacterial or viral infection manifesting as fevers or hemodynamic instability within the past 72 hours
* Lifetime cumulative daunorubicin-equivalent anthracycline dose > 368 mg/m^2
* Pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Complete remission (CR)/CR with incomplete hematologic recovery (CRi) after induction therapy | Up to day 60

SECONDARY OUTCOMES:
Proportion of patients with persistent grade 4 hematologic toxicity per Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 | At day 60
  The proportion along with the exact 95% confidence interval will reported.
Proportion of patients who achieve CR/CRi during maintenance therapy | Up to 2 years
  This is calculated only among patients who had stable disease after induction therapy and have received maintenance enasidenib monotherapy.
Proportion of patients who achieve CR/complete remission with partial hematologic recovery (CRp) after induction therapy | Up to 2 years
Time to return of normal hematopoiesis | From day 1 of induction assessed up to 2 years
  Defined as time from day 1 of induction to absolute neutrophil count (ANC) >= 1000/uL and platelet count >= 100,000/uL. The median time to return of normal hematopoiesis will be reported along with the corresponding range.
Overall survival | From day 1 of induction therapy, assessed at day 30 and 60
  Will be estimated using Kaplan-Meier methods. The survival estimate at these two time points will be reported along with a 95% confidence interval.
Proportion of patients who go on to receive allogeneic hematopoietic stem cell transplantation (HSCT) after achieving CR/CRi | Up to 2 years
  Will be reported along with an exact 95% confidence interval.

OTHER OUTCOMES:
Proportion of patients who have a particular co-occurring mutation with an allelic frequency >= 10% along with the IDH2 mutation, and have achieved CR/CRi | Up to 2 years
  Will be reported along with an exact 95% confidence interval.
Proportion of patients who achieved CR/CRi then achieve minimal residual disease negativity based on Invivoscribe assay | Up to 2 years
Proportion of abnormal troponin levels without concurrent elevated creatinine | Up to 2 years
Proportion of abnormal electrocardiogram (ECG) findings (new T-wave inversions or new ST segment abnormalities) | Up to 2 years
Proportion of echocardiogram findings with left ventricular ejection fraction reduction by >= 25% | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Caspian Oliai, MD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (3):
- United States (3):
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - University of California San Diego, San Diego, California